CLINICAL TRIAL: NCT04443829
Title: Immunotherapy Using CAR T-cells to Target CD19 for Relapsed/Refractory CD19+ Primary Central Nervous System (CNS) Lymphoma
Brief Title: Immunotherapy Using CAR T-cells to Target CD19 for Relapsed/Refractory CD19+ Primary CNS Lymphoma
Acronym: CAROUSEL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/126892
Record Dates: First submitted 2020-06-18; First posted 2020-06-23 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Primary CNS Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19CAR T-cells (Experimental): Treatment with the ATIMP: CD19CAR T-cells
  Interventions: Biological: CD19CAR T-cells

INTERVENTIONS:
Biological: CD19CAR T-cells — Infusion with: CD19CAR T-cells

SUMMARY:
The CAROUSEL Trial is a single-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product (ATIMP) in adults (age ≥16) with relapsed/refractory Primary CNS Lymphoma.

The study will evaluate the feasibility of generating the ATIMP, the safety of administering CD19CAR T-cell therapy and how effectively CD19CAR T-cells engraft, expand and persist following administration in patients with relapsed/refractory primary CNS lymphoma.

DETAILED DESCRIPTION:
The CAROUSEL Trial is a single-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product (ATIMP) in adults (age ≥16) with relapsed/refractory Primary CNS Lymphoma. The ATIMP for this study is cryopreserved autologous patient-derived T-cells transduced with CD19CAR vector to generate CD19CAR T-cells.

Patients will undergo an unstimulated leucapheresis for the generation of the ATIMP which will take approximately 15 days to generate. During this period, patients may receive "holding" chemotherapy as per institutional practice to maintain disease control. Patients will receive pre-conditioning lymphodepleting (LD) chemotherapy with cyclophosphamide 60mg/kg on Day -6, fludarabine 30mg/m2 administered over 3 days (Day -5 to Day -3) and pembrolizumab 200mg on Day -1.

All patients will be treated on Theme 1 of the study with 250 x 10^6 CD19 CAR T-cells i.v. following LD chemotherapy as described above. Patients with response of Stable Disease (SD) or Progressive Disease (PD) at Day 28 (or frank relapse beyond Day 28) and in the absence of severe toxicity related to the ATIMP, will be potentially eligible for Theme 2 of the study where they can receive Dose 2, a single dose of 25 x 10^6 CD19CAR T-cells intraventricularly via an Ommaya reservoir following LD chemotherapy as described above.

The study will evaluate the feasibility of generating the ATIMP, the safety of administering CD19CAR T-cell therapy and how effectively CD19CAR T-cells engraft, expand and persist following administration in patients with relapsed/refractory primary CNS lymphoma.

Following infusion of CD19CAR T-cell therapy patients will be monitored for between 2-4 weeks as an inpatient. Following discharge, patients will enter the interventional follow up phase and be followed up for 2 years. Patients will be seen monthly for the first 6 months, then 6 weekly to 12 months and then 3 monthly until 2 years post CD19CAR T-cell infusion.

If patients relapse within the first 2 years post CD19CAR T-cell infusion they will come off the interventional follow up and will be followed up annually until the end of trial is declared.

After completing the interventional phase of the study all patients, irrespective of whether they progressed or responded to treatment, will enter long term follow up until the end of trial is declared.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥16
2. Patients with a histologically confirmed Diffuse Large B-Cell Lymphoma (DLBCL) confined to the CNS (Primary CNS Lymphoma (PCNSL))
3. Relapsed* or refractory CD19+ PCNSL, defined as disease progression following CR/CRu/PR, or failure to achieve PR, after one or more lines of a high-dose methotrexate-containing protocol *Histological confirmation by re-biopsy at relapse is recommended if feasible. However, patients will be eligible without re-biopsy provided the initial diagnostic material is available and current MRI imaging features are consistent with PCNSL by neuroradiology review.
4. Measurable disease on contrast-enhanced MRI
5. Unsuitable for alternative salvage therapies as determined by their treating physician
6. Agreement to have a pregnancy test, use highly effective contraception (if applicable)
7. Written informed consent** ** Some patients with PCNSL may be incapable of providing their own consent due to the neurological effects of their disease. In these cases a legal representative may be sought to provide consent'.

Exclusion Criteria (Registration):

1. CD19 negative disease
2. Evidence of secondary CNS lymphoma
3. Prior allogeneic haematopoietic stem cell transplant
4. Active hepatitis B, C or HIV infection
5. Oxygen saturation ≤90% on air
6. Bilirubin >2 x upper limit of normal
7. Glomerular Filtration Rate (GFR) <50ml/min
8. Women who are pregnant or breast feeding
9. Inability to tolerate leucapheresis
10. ECOG 3-4
11. Known allergy to albumin or Dimethyl sulfoxide (DMSO)
12. Life expectancy <3months
13. Arrhythmias or significant cardiac disease and left ventricular ejection fraction <40%
14. Pre-existing neurological disorders (other than CNS involvement of underlying haematological malignancy)
15. Any contraindications to PD-1 antibody Pembrolizumab
16. History of autoimmune disease (e.g. Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 24 months
17. Evidence of active pneumonitis on chest computed tomography (CT) or positron emission tomography (PET)-CT scan at screening or history of drug-induced pneumonitis, idiopathic pulmonary fibrosis, organising pneumonia (e.g. bronchiolitis obliterans), or idiopathic pneumonitis. Prior radiation pneumonitis in the radiation field (fibrosis) is allowed (if >24 weeks since the event)

Exclusion criteria: for CD19CAR T-cell infusion ( Dose 1/i.v. and Dose 2/intraventricular):

1. Severe intercurrent infection at the time of scheduled CD19CAR T-cell infusion
2. Requirement for supplementary oxygen or active pulmonary infiltrates at the time of scheduled CD19CAR T-cell infusion
3. Theme 2 only:

   1. presence of grade 3 or 4 ICANS casually related to the ATIMP following infusion of Dose 1
   2. grade 1-2 neurotoxicity (if occurred) following Theme 1 dosing (Dose 1/i.v CD19CAR Tcell dose) that has not fully resolved prior to proposed administration of 2nd CD19CAR T-cell infusion (Dose /intraventricular) for theme 2
   3. grade 3-4 CRS following infusion of Dose 1
   4. persisting grade 2 CRS following Theme 1 dosing (Dose 1/i.v CD19CAR T-cell dose) that has not resolved to ≤ grade 1 CRS prior to proposed administration of 2nd CD19CAR Tcell infusion (Dose 2/intraventricular) for theme 2
   5. pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity evaluated by the incidence of grade 3-5 toxicity causally related to the ATIMP | 28 days
  Toxicity following CD19CAR T-cell administration as evaluated by the incidence of grade 3-5 toxicity causally related to the ATIMP
Feasibility of manufacturing CD19CAR T-cells evaluated by the number of therapeutic products generated | 28 days
  Feasibility of adequate leucapheresis collection and generation of CD19CAR T-cells as evaluated by the number of therapeutic products generated.

SECONDARY OUTCOMES:
Response at 1 and 3 months | From CD19CAR T-cells infusion to 1 and 3 months
  Proportion of patients achieving a Complete Response (CR) or Partial Response (PR) at 1 and 3 months post CD19CAR T-cells infusion: Theme 1 (i.v.) and Theme 2 (intraventricular)
Frequency of circulating CD19CAR T-cells in peripheral blood | From CD19CAR T-cells infusion up to 2 years post CD19CAR T-cells infusion
  Frequency of circulating CD19CAR T-cells in peripheral blood as assessed by flow cytometry and qPCR
Incidence of B-cell aplasia | From CD19CAR T-cells infusion up to 2 years post CD19CAR T-cells infusion
  Incidence of B-cell aplasia
Relapse rate at 1 and 2 years | At 1 year and 2 years after CD19CAR T-cells infusion
  Proportion of patients who have relapsed at 1 and 2 years after CD19CAR T-cells infusion
Progression Free Survival (PFS) at 1 and 2 years | At 1 year and 2 years after CD19CAR T-cells infusion
  Progression Free Survival at 1 and 2 years after CD19CAR T-cells infusion
Overall Survival (OS) at 1 and 2 years | At 1 year and 2 years after CD19CAR T-cells infusion
  Overall Survival at 1 and 2 years after immunotherapy with CD19CAR T-cells infusion

CONTACTS AND LOCATIONS:
Overall Officials: Claire Roddie, Study Chair — University College London Hospital
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No